CLINICAL TRIAL: NCT06675292
Title: Psychometric Properties of the Headache Needs Assessment (HANA) Survey in Tension Type Headache: Turkish Version, Reliability, and Validity Study
Brief Title: Psychometric Properties of the Turkish Version of the HANA in Tension Type Headache
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halime Arikan, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: 83116987-504
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Tension Type Headache
Keywords: Headache Needs Assessment Survey; Tension type headache; Turkish
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals with tension type headache
  Interventions: Other: Survey-based study

INTERVENTIONS:
Other: Survey-based study — The demographic information of individuals with tension-type headaches, along with data from the Visual Analog Scale, Migraine Disability Assessment Questionnaire, Headache Impact Test-6, Henry Ford Hospital Headache Disability Inventory, and Headache Needs Assessment, will be collected and analyzed.

SUMMARY:
Individuals with tension type headache

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of tension-type headache,
* Being between 18 and 65 years of age.

Exclusion Criteria:

* Having a diagnosis of any headache disorder other than tension-type headache,
* Having a history of any systemic disease, such as malignancy, inflammatory conditions, acute fractures, surgical history, or neurological, psychological, or rheumatological disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with tension type headache
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Headache Needs Assessment Survey | through study completion, an average of 1 month
  The Headache Needs Assessment consists of seven items that evaluate areas such as anxiety/worry, depression/discouragement, self-control, energy, functioning/work, family/social activities, and the overall impact of migraine. A unique aspect of the questionnaire is that it separates responses into two categories: (1) How often did this issue occur? (1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Always); and (2) How much did this issue bother you? (1 = Not at all, 2 = A little, 3 = Somewhat, 4 = A lot, 5 = Very much). The total score ranges from 14 to 70, with higher scores indicating a greater negative impact on quality of life.

SECONDARY OUTCOMES:
Visual Analog Scale | through study completion, an average of 1 month
  Headache severity will be assessed using the Visual Analog Scale (VAS). For the VAS, a 10 cm horizontal line is drawn with a ruler. The beginning of the line (0 cm) is described to patients as "no pain," and the end of the line (10 cm) as "unbearable, severe pain." Patients are asked to mark a point on the line that best represents the intensity of their headache between these two endpoints. The distance from the starting point to the marked location is then measured and recorded as the headache severity.
Headache Impact Test-6 (HIT-6) | through study completion, an average of 1 month
  Headache Impact Test-6 (HIT-6), a quality of life questionnaire for headaches that assesses vitality, pain, psychological distress, social functioning, role limitations, and cognitive functioning. Each item is scored on a 5-point Likert scale (6 = never, 8 = rarely, 10 = sometimes, 11 = very often, 13 = always). The total score is calculated by summing the scores of all six items, ranging from 36 to 78. Scores are categorized as follows: ≤49 = little to no impact, 50-55 = some impact, 56-59 = substantial impact, and 60-78 = severe impact, with higher scores indicating greater impairment in quality of life. The validity, reliability, and Turkish version of the questionnaire have been established.
Henry Ford Hospital Headache Disability Inventory | through study completion, an average of 1 month
  The Henry Ford Hospital Headache Disability Inventory is a 25-item questionnaire designed to assess the impact of headaches on daily life. This inventory has a two-dimensional structure, comprising emotional and functional components. Items are scored as No: 0, Sometimes: 2, and Yes: 4. The total score ranges from 0 to 100, with higher scores indicating greater headache-related disability. The validity, reliability, and Turkish version of the inventory have been established by Kılınç et al.

CONTACTS AND LOCATIONS:
Overall Officials: Halime ARIKAN, Doctor of Philosophy, Principal Investigator — Tokat Gaziosmanpaşa University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

REFERENCES:
- [Derived] Arikan H, Onan D, Kulu U. Psychometric properties of the headache needs assessment (HANA) survey in tension type headache: Turkish version, reliability, and validity study. Acta Neurol Belg. 2025 Aug;125(4):1091-1099. doi: 10.1007/s13760-025-02749-4. Epub 2025 Feb 24. PMID 39992579